CLINICAL TRIAL: NCT02367573
Title: 3D Versus 2D HD Laparoscopy in Inguinal Hernia Repair: a Prospective, Single Blinded, Randomized, Controlled Trial
Brief Title: 3D vs 2D HD Laparoscopy in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Koppatz, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUCH-328-150128
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 2D TAPP (Active Comparator): Trans-abdominal pre-peritoneal laparoscopic inguinal hernia repair operated with two dimensional view
  Interventions: Procedure: 2D laparoscopic TAPP inguinal hernia repair
- 3D TAPP (Experimental): Trans-abdominal pre-peritoneal laparoscopic inguinal hernia repair operated with three dimensional view
  Interventions: Procedure: 3D laparoscopic TAPP inguinal hernia repair

INTERVENTIONS:
Procedure: 2D laparoscopic TAPP inguinal hernia repair
  Arms: 2D TAPP
Procedure: 3D laparoscopic TAPP inguinal hernia repair
  Arms: 3D TAPP

SUMMARY:
Inguinal hernia can be repaired laparoscopically. In the normal laparoscopy there are only two-dimensional view, which is somewhat challenging when operating in three-dimensional environment. The three-dimensional laparoscopic systems are gradually entering the operating rooms. There are plenty of evidence of the benefits of 3D-system in laboratory conditions. However, no prospective randomized trials have been published in the clinical point of view. Therefore, the purpose of this study is to investigate is there something to gain in changing into 3D laparoscopic system in the transabdominal pre-peritoneal (TAPP) inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic inguinal hernia repair

Exclusion Criteria:

* Some other surgical operation planned during TAPP
* Expected major risk of conversion (e.g. multiple previous abdominal operation, previous peritonitis)
* Operating surgeon experience less than 5 3D laparoscopy operations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Duration of surgery | Expected average time of surgery 1 hour

SECONDARY OUTCOMES:
Need for conversion into open surgery | During the operation, expected average time of surgery 1 hour
Intraoperative complications | During the operation, expected average time of surgery 1 hour
  Any complication during the operation e.g. hemorrhagic, intestine or bladder rupture
Complications, Clavien-Dindo classification | 30 days after randomization
Postoperative stay in hospital | Expected range 0-7 day
Bleeding | During the operation, expected average time of surgery 1 hour
Number of participants with readmission(s) | 30 days after randomization
Total need of opioids in milligrams | Expected range 0-7 day
Mortality | 30 days after randomization
Operation theatre time | Expected average 1,5 hours
Postoperative pain, VAS | Expected range 0-7 day

OTHER OUTCOMES:
Incisional hernias | after 1, 5 and 10 year
Inguinal hernia recurrence | after 1, 5 and 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, MD,PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Koppatz HE, Harju JI, Siren JE, Mentula PJ, Scheinin TM, Sallinen VJ. Three-dimensional versus two-dimensional high-definition laparoscopy in transabdominal preperitoneal inguinal hernia repair: a prospective randomized controlled study. Surg Endosc. 2020 Nov;34(11):4857-4865. doi: 10.1007/s00464-019-07266-z. Epub 2019 Nov 21. PMID 31754852